CLINICAL TRIAL: NCT05683132
Title: Increasing PTSD Treatment Engagement in Women Veterans: Role of CBT for Insomnia (CDA 20-227)
Brief Title: Treatments in Women Veterans With Insomnia and PTSD
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: VA Office of Research and Development (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CDX 22-009
Record Dates: First submitted 2022-12-21; First posted 2023-01-12 (Actual); Last update posted 2026-01-05 (Actual); Status verified 2025-12

CONDITIONS: Insomnia; PTSD; Women Veterans
Keywords: Insomnia Disorder; Posttraumatic Stress Disorder; Women's Health
MeSH Terms: conditions — Sleep Initiation and Maintenance Disorders; Stress Disorders, Post-Traumatic

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Masking Description: Outcome assessors will be blinded from group assignment and the treatment content. Participants will be blinded to the content of the treatment arm to which they are not assigned.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Trauma-Informed CBT-I (Experimental): This intervention includes trauma-informed adaptations to standard treatment for insomnia, CBT-I
  Interventions: Behavioral: Trauma-Informed CBT-I
- PTSD Psychoeducation (Active Comparator): This intervention includes psychoeducation about PTSD symptoms modeled after usual care in a VA Women's Health Clinic.
  Interventions: Behavioral: PTSD Psychoeducation

INTERVENTIONS:
Behavioral: Trauma-Informed CBT-I — 5 individual sessions incorporating behavioral and cognitive therapy components and trauma-informed adaptations with a trained instructor.
  Arms: Trauma-Informed CBT-I
Behavioral: PTSD Psychoeducation — 5 individual sessions incorporating psychoeducation about PTSD symptoms with a trained instructor.
  Arms: PTSD Psychoeducation

SUMMARY:
This pilot trial will compare trauma-informed Cognitive Behavioral Therapy for Insomnia (CBT-I) to a psychoeducational intervention in women Veterans with comorbid insomnia and posttraumatic stress disorder (PTSD). The CBT-I intervention includes trauma-informed adaptations to an insomnia treatment and the psychoeducational intervention is modeled after usual care in a VA Women's Mental Health Clinic.

The study objectives are to: 1) Iteratively refine the structure and materials of trauma-informed CBT-I in preparation for a pilot trial, 2) Pilot test the effects of trauma-informed CBT-I on PTSD treatment readiness and engagement in a sample of women Veterans, and 3) Examine potential mechanisms underlying variations in PTSD treatment readiness and engagement over time among women Veterans.

Women Veterans with insomnia and comorbid PTSD who receive care at Sepulveda and West Los Angeles facilities will be recruited for the study. Those who pass an initial eligibility screen will be enrolled and written informed consent will be obtained. A baseline assessment will be completed that includes measures of PTSD treatment readiness, perceived barriers to PTSD treatment, and sleep and mental health symptoms. Then Veterans who meet all eligibility criteria will be randomly assigned to trauma-informed CBT-I (n=25) or the psychoeducational intervention (n=25). Both treatments will be provided in 5 one-on-one sessions by a trained instructor who is supervised by a behavioral sleep medicine specialist. All randomized participants (n=50) will have 2 follow-up assessments (post-treatment and 3-months). The follow-up assessments will collect information on PTSD treatment readiness, perceived barriers to PTSD treatment, and sleep and mental health symptoms. Chart reviews will be conducted 6-months post-treatment to assess number of PTSD treatment appointments attended (treatment engagement measure). Qualitative interviews will be conducted to identify mechanisms underlying PTSD treatment engagement.

DETAILED DESCRIPTION:
Posttraumatic stress disorder (PTSD) is the most common psychiatric service-connected condition among women Veterans, yet many women Veterans do not receive evidence-based psychotherapies for PTSD. PTSD and insomnia disorder are highly comorbid in women Veterans and research suggests that insomnia is a risk factor for PTSD development and severity, while healthy sleep is associated with improved mood, daytime functioning, enhanced learning, and increased emotion regulation. Addressing insomnia symptoms in women Veterans may offer an early point of intervention to reduce insomnia and some PTSD symptoms, while also providing a novel approach to improve patient engagement in PTSD treatments. No previous studies have examined the impact of trauma-informed Cognitive Behavioral Therapy for insomnia (CBT-I) on sleep and psychiatric symptoms among women Veterans with comorbid insomnia disorder and PTSD.

This pilot trial will compare trauma-informed CBT-I to a psychoeducational intervention in women Veterans with comorbid insomnia and PTSD. The CBT-I intervention includes trauma-informed adaptations to an insomnia treatment and the psychoeducational intervention is modeled after usual care in a VA Women's Mental Health Clinic.

The study objectives are to: 1) Iteratively refine the structure and materials of trauma-informed CBT-I in preparation for a pilot trial, 2) Pilot test the effects of trauma-informed CBT-I on PTSD treatment readiness and engagement in a sample of women Veterans, and 3) Examine potential mechanisms underlying variations in PTSD treatment readiness and engagement over time among women Veterans.

Women Veterans with insomnia and comorbid PTSD who receive care at Sepulveda and West Los Angeles facilities will be recruited for the study. Those who pass an initial eligibility screen will be enrolled and written informed consent will be obtained. A baseline assessment will be completed that includes measures of PTSD treatment readiness, perceived barriers to PTSD treatment, and sleep and mental health symptoms. The first 5 eligible participants will receive trauma-informed CBT-I and provide feedback to guide intervention refinement. Then Veterans who meet all eligibility criteria will be randomly assigned to trauma-informed CBT-I (n=25) or the psychoeducational intervention (n=25). Both treatments will be provided in 5 one-on-one sessions by a trained instructor who is supervised by a behavioral sleep medicine specialist. All randomized participants (n=50) will have 2 follow-up assessments (post-treatment and 3-months). The follow-up assessments will collect information on PTSD treatment readiness, perceived barriers to PTSD treatment, and sleep and mental health symptoms. A chart review will be conducted 6-months post-treatment to assess number of PTSD treatment appointments attended (i.e., treatment engagement measure). Qualitative interviews (n=20) will be conducted with pilot completers and non-completers to identifying other facilitators of and barriers to PTSD treatment engagement.

ELIGIBILITY:
Inclusion Criteria:

* Community-dwelling women Veterans aged 18 years and older
* Received care from VAGLAHS
* Have symptoms of PTSD
* Have symptoms of insomnia

Exclusion Criteria:

* Reported health or emotional problems, or use of drugs or alcohol that would make it difficult for them to participate in this study
* Too ill to engage in the study procedures
* Unable to self-consent to participate
* Previously engaged in Cognitive Behavioral Therapy for Insomnia (CBT-I) treatment
* Previously engaged in PTSD psychoeducational group offered in VAGLAHS Women's Health Clinic
* Previously completed >3 sessions of PTSD treatment (Cognitive Processing Therapy and/or Prolonged Exposure)
* Pregnant or pregnant within 6 months of study
* Untreated moderate to severe obstructive sleep apnea diagnosis as evidenced by Apnea Hypopnea Index (AHI) in chart and/or screens that indicate high risk
* Unstable housing
* Inability to read, write, and communicate in English
* Unstable medical or psychiatric disorders (which is a contraindication for behavioral treatment of insomnia)
* Remission of PTSD or insomnia symptoms

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Only women Veterans will be eligible for the study.
Enrollment: 100 (Estimated)
Dates: Start 2023-06-01 (Actual); Primary Completion 2027-12-31 (Estimated); Study Completion 2028-12-31 (Estimated)

PRIMARY OUTCOMES:
University of Rhode Island Change Assessment Scale (URICA) | Post-Treatment (approximately 1 week after last intervention session)
  The problem-specific URICA (psychotherapy version) is a 32-item questionnaire that assesses respondent's readiness to change at entrance to treatment. The URICA includes 4 subscales measuring the stages of change: Precontemplation (P), Contemplation (C), Action (A), and Maintenance (M). To obtain a readiness to change score, first sum items from each subscale and divide by 7 to get the mean for each subscale. One item from each subscale is omitted for the subscale mean calculations for the 32-item version of the URICA (items 4, 9, 20, and 31). Then sum the means from the Contemplation, Action, and Maintenance subscales and subtract the Precontemplation mean (C + A + M - PC = Readiness). Scores range from -2 to 14. Higher scores will indicate greater readiness.
Readiness for Psychotherapy Index (RPI) | Post-Treatment (approximately 1 week after last intervention session)
  The RPI is a 20-item questionnaire that assesses respondent's readiness to engage in psychotherapy. The RPI consists of 4 subscales including: disinterest, perseverance, openness, and distress. To obtain a readiness score, sum items from each subscale. Then sum the scores from the perseverance, openness, and distress subscales and subtract the disinterest subscale score (Perseverance + Openness + Distress - Disinterest = Readiness). Scores range from -10 to 70. Higher scores will indicate greater readiness.
University of Rhode Island Change Assessment Scale (URICA) | 3-month Follow-up (approximately 90 days after last intervention session)
  The problem-specific URICA (psychotherapy version) is a 32-item questionnaire that assesses respondent's readiness to change at entrance to treatment. The URICA includes 4 subscales measuring the stages of change: Precontemplation (P), Contemplation (C), Action (A), and Maintenance (M). To obtain a readiness to change score, first sum items from each subscale and divide by 7 to get the mean for each subscale. One item from each subscale is omitted for the subscale mean calculations for the 32-item version of the URICA (items 4, 9, 20, and 31). Then sum the means from the Contemplation, Action, and Maintenance subscales and subtract the Precontemplation mean (C + A + M - PC = Readiness). Scores range from -2 to 14. Higher scores will indicate greater readiness.
Readiness for Psychotherapy Index (RPI) | 3-month Follow-up (approximately 90 days after last intervention session)
  The RPI is a 20-item questionnaire that assesses respondent's readiness to engage in psychotherapy. The RPI consists of 4 subscales including: disinterest, perseverance, openness, and distress. To obtain a readiness score, sum items from each subscale. Then sum the scores from the perseverance, openness, and distress subscales and subtract the disinterest subscale score (Perseverance + Openness + Distress - Disinterest = Readiness). Scores range from -10 to 70. Higher scores will indicate greater readiness.
Frequency of PTSD Treatment Appointments | 6-month Follow-up (180 days after last intervention session)
  A structured medical record review will be performed 6 months post-treatment to obtain information on utilization of VA healthcare services during the time period between the last intervention session and 180 days after the last intervention session. Reviews will identify the presence and frequency of mental health appointments with evidence-based practice (EBP) health codes and/or Cognitive Processing Therapy (CPT) and Prolonged Exposure (PE) note templates, which are psychotherapies to treat PTSD. Attendance will be measured as a count, ranging from 0 to an unlimited value. Higher counts will indicate greater engagement in PTSD treatment.

CONTACTS AND LOCATIONS:
Overall Officials: Gwendolyn C Carlson, PhD, Principal Investigator — VA Greater Los Angeles Healthcare System, West Los Angeles, CA
Locations (1):
- VA Greater Los Angeles Healthcare System, West Los Angeles, CA, West Los Angeles, California, United States

IPD SHARING:
Plan to Share IPD: No